CLINICAL TRIAL: NCT00508833
Title: Safety and the Efficacy of GSK Biologicals' Candidate Adjuvanted Vaccines (287615) Containing HBsAg With Various Adjuvants to Induce Cytotoxic T Lymphocytes (CTL) in Healthy Adult Volunteers
Brief Title: Safety and Efficacy of SmithKline Beecham (GlaxoSmithKline [GSK]) Biologicals' Candidate Adjuvanted Vaccines (287615)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 287615/005
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2007-07-30 (Estimated); Status verified 2007-07

CONDITIONS: Hepatitis B Disease
Keywords: Adjuvants; HBsAg

INTERVENTIONS:
Biological: 287615 containing HBsAg with adjuvants

SUMMARY:
This study was done to evaluate the effect of various adjuvants in combination with HBsAg as a model antigen on the induction of immune responses, mainly cytotoxic T lymphocytes (CTL) in healthy volunteers. The study was also done to evaluate the safety and reactogenicity of the various adjuvanted vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 40 years of age
* Written informed consent obtained from subject
* Female of non-childbearing potential

Exclusion Criteria:

* Any hepatitis B vaccination.
* Positive HBV serological markers: anti-HBs, anti-HBc, and/ or HBsAg
* Pregnancy or lactating female
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days or 7 half-lives (whichever is the longer) preceding the first vaccine administration

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2000-03

PRIMARY OUTCOMES:
Intensity of the CTL response at Week 6

SECONDARY OUTCOMES:
Solicited symptoms (7 days), other AEs (up to 6 mths), SAEs (entire study), intensity of CTL response at Week 46, 48, 78; anti-HBs response up to week 78

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Ghent, Belgium